CLINICAL TRIAL: NCT05208203
Title: Acute Ischemic Stroke "Green Channel" Registry--Xuanwu Hospital
Brief Title: XuanwuH Acute Ischemic Stroke Registry
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, qingfengma, MD, Xuanwu Hospital, Beijing
Other Study IDs: qingfeng ma stroke xuanwuH
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Cerebrovascular disease
MeSH Terms: conditions — Ischemic Stroke; Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke patients: acute ischemic stroke patients including all treatments.
  Interventions: Other: telephone call d90

INTERVENTIONS:
Other: telephone call d90 — telephone call on day 90 to assess the primary outcome (mRs d90)

SUMMARY:
Acute ischemic stroke registry--Xuanwu Hospital(XSR) is an academic, independent, prospective, single center, observational registry study. Consecutive acute ischemic stroke patients assessed in stroke "green channel" of Xuanwu Hospital(China) will be enrolled in our study. Patients receive regular treatment and data will be collected as part of clinical routine. Baseline clinical and procedural information as well clinical follow-up information during in-hospital stay, and up to 90 days of stroke onset are collected. Data collected include demographics, National Institute of Health Stroke Scale (NIHSS) on admission, pre-treatment ASPECTS, information on timing and success of thrombolysis or thrombectomy, procedural complications, intracranial hemorrhage, and functional outcome.The study aim to investigate the real situation of assessment, diagnosis and treatment of acute ischemic stroke patients in "green channel",and verify the effect of the improvement of "green channel" process in the diagnosis and treatment of patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke or transient ischemic attack(TIA)
* Age >18 years
* Ethic approval in process
* Receiving assessment in stroke "green channel" of Xuanwu Hospital

Exclusion Criteria:

* Non-acute ischemic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all acute stroke patients with the clinical diagnosis of acute ischemic stroke, Age >18 years
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
modified ranking scale on day (mRs) day 90 | 90 days
  mRs: modified ranking scale; the scale is a commonly used measurement for the degree of disability or dependence in the daily activities of people who have suffered a stroke; scale range 0-6, with 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms. 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.

SECONDARY OUTCOMES:
Stroke Event | 1year
  The patients were monitored whether they recured ischemic stroke event including transient ischemic attack (TIA) or stroke confirmed by neurologist and diffusion-weighted image MRI.
adverse event | 1year
  The patients were monitored whether they appeared symptomatic intracranial hemorrhage,cerebral hernia or other life-threatening events.

CONTACTS AND LOCATIONS:
Overall Officials: qingfeng Ma, MD, Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] GBD 2016 Neurology Collaborators. Global, regional, and national burden of neurological disorders, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):459-480. doi: 10.1016/S1474-4422(18)30499-X. Epub 2019 Mar 14. PMID 30879893
- [Background] Harris D, Hall C, Lobay K, McRae A, Monroe T, Perry JJ, Shearing A, Wollam G, Goddard T, Lang E. Canadian Association of Emergency Physicians position statement on acute ischemic stroke. CJEM. 2015 Mar;17(2):217-26. doi: 10.1017/cem.2015.26. PMID 26120643
- [Result] van Swieten JC, Koudstaal PJ, Visser MC, Schouten HJ, van Gijn J. Interobserver agreement for the assessment of handicap in stroke patients. Stroke. 1988 May;19(5):604-7. doi: 10.1161/01.str.19.5.604. PMID 3363593